CLINICAL TRIAL: NCT00296192
Title: A Double-Blind, Placebo-Controlled, Parallel-Group, Proof of Concept Trial to Assess the Tolerability, Safety, and Efficacy of Rotigotine Nasal Spray for the Acute Treatment of "OFF" Symptoms in Subjects With Advanced-Stage, Idiopathic Parkinson Disease
Brief Title: Efficacy, Safety and Tolerability of Rotigotine Nasal Spray for the Acute Treatment of Parkinson Symptoms
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SP0873; EudraCT: 2005-004290-19 (Other: EudraCT)
Record Dates: First submitted 2006-02-22; First posted 2006-02-24 (Estimated); Results first posted 2010-01-29 (Estimated); Last update posted 2014-10-02 (Estimated); Status verified 2011-02

CONDITIONS: Parkinson's Disease
Keywords: Rotigotine; Rotigotine nasal spray; Efficacy, safety and tolerability; Parkinson's disease
MeSH Terms: conditions — Parkinson Disease | interventions — rotigotine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Placebo 1 (Placebo Comparator): Placebo nasal spray 1 - 4 puffs
  Interventions: Other: Placebo
- Rotigotine 1 (Experimental): Rotigotine Nasal Spray 1 puff (0.25 mg Rotigotine)
  Interventions: Drug: Rotigotine nasal spray
- Rotigotine 2 (Experimental): Rotigotine Nasal Spray - 2 puffs (0.49 mg Rotigotine)
  Interventions: Drug: Rotigotine nasal spray
- Rotigotine 3 (Experimental): Rotigotine Nasal Spray - 3 puffs (0.74 mg Rotigotine)
  Interventions: Drug: Rotigotine nasal spray
- Rotigotine 4 (Experimental): Rotigotine Nasal Spray - 4 puffs (0.99 mg Rotigotine)
  Interventions: Drug: Rotigotine nasal spray

INTERVENTIONS:
Drug: Rotigotine nasal spray — Rotigotine- HCl 2.5mg/mL nasal spray, dosage per puff of 275µg per 110µg administered in up to 4 deliveries
  Other Names: Neupro; SPM 952
  Arms: Rotigotine 1; Rotigotine 2; Rotigotine 3; Rotigotine 4
Other: Placebo — placebo nasal spray 1, 2 3, and 4 puffs
  Arms: Placebo 1

SUMMARY:
The objective of this trial is to evaluate safety and efficacy of rotigotine nasal spray (SPM 952) in a single dose application scheme.

Subjects will undergo a 2 - 28 days screening period in which eligibility criteria will be checked. Subjects will then be hospitalized for one night. In the morning of the next day, subjects will be randomly assigned either to rotigotine or placebo nasal spray and will then receive a single dose of trial medication. Safety assessments after application include adverse events, 12-lead electrocardiograms, blood pressure and heart rate assessments, and laboratory checks. Efficacy will be assessed by application of motor examination scores.

The first subject is planned to be enrolled in February 2006. The last subject is planned to be enrolled in May 2006. Last subject out is expected for August 2006.

DETAILED DESCRIPTION:
The objective of this trial is to evaluate safety and efficacy of rotigotine nasal spray (SPM 952)in a single dose application scheme. Subjects will undergo a 2-28 days screening period in which eligibility criteria will be checked. Subjects will then be hospitalized for one night. In the morning of the next day, subjects will be randomly assigned either to rotigotine or placebo nasal spray and will then receive a single dose of trial medication. Safety assessments after application include adverse events, 12-lead electrocardiograms, blood pressure and heart rate assessments, and laboratory checks. Efficacy will be assessed by application of motor examination scores.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects with idiopathic Parkinson's disease for at least 3 years in duration
* At least 30 years of age

Exclusion Criteria:

* Patients with atypical Parkinson's or clinically relevant concomitant diseases or medical conditions

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2006-02; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants flow shows all subjects randomized. Safety analyses are based on actual treatment received; 4 subjects randomized to placebo were mistreated (1 subject each in the rotigotine 1 puff, rotigotine 2 puffs, rotigotine 3 puffs, and rotigotine 4 puffs treatment arms).
Groups:
- Placebo 1-4 Puffs: Placebo nasal spray 1 - 4 puffs
- Rotigotine 1 Puff: Rotigotine Nasal Spray 1 puff (0.25 mg Rotigotine)
- Rotigotine 2 Puffs: Rotigotine Nasal Spray - 2 puffs (0.49 mg Rotigotine)
- Rotigotine 3 Puffs: Rotigotine Nasal Spray - 3 puffs (0.74 mg Rotigotine)
- Rotigotine 4 Puffs: Rotigotine Nasal Spray - 4 puffs (0.99 mg Rotigotine)
Period: Overall Study
Arm/Group | Placebo 1-4 Puffs | Rotigotine 1 Puff | Rotigotine 2 Puffs | Rotigotine 3 Puffs | Rotigotine 4 Puffs
Started | 17 | 16 | 16 | 17 | 16
Completed | 17 | 16 | 16 | 17 | 16
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo 1-4 Puffs | Rotigotine 1 Puff | Rotigotine 2 Puffs | Rotigotine 3 Puffs | Rotigotine 4 Puffs | Total
Number analyzed (Participants) | 17 | 16 | 16 | 17 | 16 | 82
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 8 | 5 | 9 | 10 | 41
  >=65 years | 8 | 8 | 11 | 8 | 6 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.9 (6.94) | 67.1 (7.54) | 66.8 (9.67) | 63.9 (8.28) | 60.5 (8.04) | 64.4 (8.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 4 | 7 | 4 | 24
  Male | 13 | 11 | 12 | 10 | 12 | 58
Region of Enrollment [Number; unit: participants]
  Germany | 11 | 12 | 12 | 10 | 13 | 58
  Austria | 2 | 2 | 1 | 4 | 1 | 10
  United Kingdom | 1 | 1 | 2 | 0 | 2 | 6
  Spain | 3 | 1 | 1 | 3 | 0 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Who Complete the Trial
Time Frame: 15 days
Population: Full Analysis Set: Subjects receiving at least one delivery of trial medication and with at least one post-baseline efficacy measurement.
Measure: Number; unit: participants
Arm/Group | Placebo 1-4 Puffs | Rotigotine 1 Puff | Rotigotine 2 Puffs | Rotigotine 3 Puffs | Rotigotine 4 Puffs
Number analyzed (Participants) | 17 | 16 | 16 | 17 | 16
participants | 17 | 16 | 16 | 17 | 16

2. Secondary Outcome: Change From Baseline at 24 Minutes Post-dose in Unified Parkinson Disease Rating Scale (UPDRS) Part III Motor Examination
Description: The Unified Parkinson's Disease Rating Scale (UPDRS) is a scale for the assessment of function in Parkinson's disease. UPDRS Part III measures Motor Examination. Range: 0 (Best score possible) to 56 (Worst score possible) Change = 24 minute value minus baseline value.
Time Frame: Baseline, and 24 minutes post-dose
Population: Full Analysis Set: Subjects receiving at least one delivery of trial medication and with at least one post-baseline efficacy measurement. Missing values at 24 minutes post-dose timepoint were not imputed; number of observations at 24 minutes post-dose timepoint may be less than that for baseline timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo 1-4 Puffs | Rotigotine 1 Puff | Rotigotine 2 Puffs | Rotigotine 3 Puffs | Rotigotine 4 Puffs
Number analyzed (Participants) | 17 | 16 | 16 | 17 | 16
score on a scale
  Baseline | 35.1 (7.77) | 37.2 (10.68) | 39.5 (12.94) | 36.2 (7.60) | 37.6 (9.30)
  24 minutes post-dose | 25.3 (12.44) | 30.0 (11.35) | 29.2 (13.53) | 29.1 (8.51) | 26.4 (12.95)
  Change from baseline to 24 minutes post-dose | -9.8 (7.8) | -7.2 (10.32) | -10.3 (6.17) | -7.1 (6.47) | -11.6 (10.65)
Statistical Analysis 1: Comparison: Placebo 1-4 Puffs vs Rotigotine 1 Puff; Analysis of covariance modeling change from baseline at 24 minutes post-dose in UPDRS Part III, controlling for treatment group and baseline value; Test type: Superiority or Other; ANCOVA; Mean Difference (Net) = 2.9, 95% CI [-2.9 to 8.7], Standard Error of Mean 2.91
Statistical Analysis 2: Comparison: Placebo 1-4 Puffs vs Rotigotine 2 Puffs; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; ANCOVA; Mean Difference (Net) = 0.1, 95% CI [-5.7 to 6.0], Standard Error of Mean 2.93
Statistical Analysis 3: Comparison: Placebo 1-4 Puffs vs Rotigotine 3 Puffs; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; ANCOVA; Mean Difference (Net) = 2.9, 95% CI [-2.8 to 8.6], Standard Error of Mean 2.86
Statistical Analysis 4: Comparison: Placebo 1-4 Puffs vs Rotigotine 4 Puffs; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; ANCOVA; Mean Difference (Net) = -1.4, 95% CI [-7.4 to 4.6], Standard Error of Mean 3.02

3. Secondary Outcome: Change From Baseline to 34 Minutes Post-dose in Tapping Rate (Taps/Min)
Description: One-minute tapping rate will be calculated as the number of times a subject could tap on two 4 x 4 cm marks placed on a board 30 cm apart during 1 minute (30 cm measured from the inner border of the two boxes).
Time Frame: Baseline and 34 minutes post-dose
Population: Full Analysis Set: Subjects receiving at least one delivery of trial medication and with at least one post-baseline efficacy measurement. Missing values at 34 minutes post-dose timepoint were not imputed; number of observations at 34 minutes post-dose timepoint may be less than that for baseline timepoint.
Measure: Mean (Standard Deviation); unit: taps per minute
Arm/Group | Placebo 1-4 Puffs | Rotigotine 1 Puff | Rotigotine 2 Puffs | Rotigotine 3 Puffs | Rotigotine 4 Puffs
Number analyzed (Participants) | 17 | 16 | 16 | 17 | 16
taps per minute
  Baseline | 112.7 (47.08) | 109.8 (28.94) | 127.2 (44.33) | 115.9 (41.05) | 118.3 (40.41)
  34 minutes post-dose | 141.2 (50.92) | 131.0 (30.01) | 138.7 (44.42) | 142.9 (51.20) | 144.4 (57.64)
  Change from baseline to 34 minutes post-dose | 28.5 (27.83) | 21.2 (26.69) | 11.5 (11.27) | 27.1 (25.25) | 22.9 (27.75)
Statistical Analysis 1: Comparison: Placebo 1-4 Puffs vs Rotigotine 1 Puff; Analysis of covariance modeling change from baseline to 34 minutes post-dose in tapping rate, controlling for treatment group and baseline value; Test type: Superiority or Other; ANCOVA; Mean Difference (Net) = -8.6, 95% CI [-25.7 to 8.5], Standard Error of Mean 8.58
Statistical Analysis 2: Comparison: Placebo 1-4 Puffs vs Rotigotine 2 Puffs; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; ANCOVA; Mean Difference (Net) = -16.8, 95% CI [-34.0 to 0.4], Standard Error of Mean 8.63
Statistical Analysis 3: Comparison: Placebo 1-4 Puffs vs Rotigotine 3 Puffs; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; ANCOVA; Mean Difference (Net) = -1.4, 95% CI [-18.2 to 15.4], Standard Error of Mean 8.45
Statistical Analysis 4: Comparison: Placebo 1-4 Puffs vs Rotigotine 4 Puffs; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; ANCOVA; Mean Difference (Net) = -5.5, 95% CI [-23.3 to 12.2], Standard Error of Mean 8.90

4. Secondary Outcome: "Success Rate" (Percentage of Subjects Achieving "Off" Reversals)
Description: Subjects reversing from "off" to "on" following initiation of treatment. "On" and "off" state refer to periods where Parkinson's disease symptoms are not present ("on") and periods where symptoms are present ("off"); the "on"/"off" determination at each assessment timepoint was made by the investigator.
Time Frame: Up to 6 hours post-dose
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo 1-4 Puffs | Rotigotine 1 Puff | Rotigotine 2 Puffs | Rotigotine 3 Puffs | Rotigotine 4 Puffs
Number analyzed (Participants) | 17 | 16 | 16 | 17 | 16
percentage of participants
  Reversed from "off" to "on" (success) | 70.6 | 50.0 | 75.0 | 70.6 | 75.0
  Did not reverse from "off" to "on" | 29.4 | 50.0 | 25.0 | 29.4 | 25.0
Statistical Analysis 1: Comparison: Placebo 1-4 Puffs vs Rotigotine 1 Puff; 95% confidence interval in difference in success rate; Test type: Superiority or Other; Confidence interval; Difference in proportions = -20.6, 95% CI [-53.3 to 12.1]
Statistical Analysis 2: Comparison: Placebo 1-4 Puffs vs Rotigotine 2 Puffs; 95% confidence interval in difference in success rate; Test type: Superiority or Other; 95% confidence interval; Difference in proportions = 4.4, 95% CI [-25.9 to 34.7]
Statistical Analysis 3: Comparison: Placebo 1-4 Puffs vs Rotigotine 3 Puffs; 95% confidence interval in difference in success rate; Test type: Superiority or Other; 95% confidence interval; Difference in proportions = 0.0, 95% CI [-30.6 to 30.6]
Statistical Analysis 4: Comparison: Placebo 1-4 Puffs vs Rotigotine 4 Puffs; 95% confidence interval in difference in success rate; Test type: Superiority or Other; 95% confidence interval; Difference in proportions = 4.4, 95% CI [-25.9 to 34.7]

5. Secondary Outcome: Time of First "Off" Reversal
Description: Number of minutes to first reversal of symptoms from "off" to "on". Estimated via Kaplan-Meier estimation method. "On" and "off" state refer to periods where Parkinson's disease symptoms are not present ("on") and periods where symptoms are present ("off"); the "on"/"off" determination at each assessment timepoint was made by the investigator.
Time Frame: Up to 6 hours post-dose
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Placebo 1-4 Puffs | Rotigotine 1 Puff | Rotigotine 2 Puffs | Rotigotine 3 Puffs | Rotigotine 4 Puffs
Number analyzed (Participants) | 17 | 16 | 16 | 17 | 16
minutes | 50 [24 to 65] | 60 [40 to 60] | 51 [22 to 84] | 50 [35 to 70] | 59 [35 to 190]

ADVERSE EVENTS:
Description: Safety analyses are based on actual treatment received; 4 subjects randomized to placebo were mistreated (1 subject each in the rotigotine 1 puff, rotigotine 2 puffs, rotigotine 3 puffs, and rotigotine 4 puffs treatment arms).
Arm/Group | Placebo 1-4 Puffs | Rotigotine 1 Puff | Rotigotine 2 Puffs | Rotigotine 3 Puffs | Rotigotine 4 Puffs
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/17 | 1/17 | 0/18 | 1/17
Other Adverse Events (participants affected / at risk) | 3/13 | 9/17 | 5/17 | 9/18 | 9/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo 1-4 Puffs (N=13) | Rotigotine 1 Puff (N=17) | Rotigotine 2 Puffs (N=17) | Rotigotine 3 Puffs (N=18) | Rotigotine 4 Puffs (N=17)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo 1-4 Puffs (N=13) | Rotigotine 1 Puff (N=17) | Rotigotine 2 Puffs (N=17) | Rotigotine 3 Puffs (N=18) | Rotigotine 4 Puffs (N=17)
Atrioventricular block first degree (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (6)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Salivary hypersecretion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Application site reaction (General disorders) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 2 (2)
Application site irritation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Application site dryness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Application site paraesthesia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Difficulty in walking (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Blood urine present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
White blood cells urine (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
White blood cells urine postitive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
Somnolence (Nervous system disorders) | 1 (1) | 2 (2) | 2 (2) | 3 (3) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dystonia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Burning sensation (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokinesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sleep attacks (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Yawning (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pallor (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
UCB has > 60 days but <= 180 days to review results communications prior to public release and may delete information that is confidential and compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.